CLINICAL TRIAL: NCT03233659
Title: Study of the Function of Immune System in Patients Undergoing Allogeneic Stem Cell Transplantation
Brief Title: Immune Monitoring After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Mario Arpinati, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: IMM-2011-01
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Allogeneic Stem Cell Transplantation; GVHD
Keywords: Allogeneic Stem Cell Transplantation, APCs, GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of serum and PBMC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BMT patients: All patients undergoing Allogeneic Stem Cell Transplantation are enrolled in the study.

SUMMARY:
Graft versus Host disease ( GVHD) is one of the major complications of Allogeneic Stem Cell Transplantation. Acute GVHD develops early ( within 2to 3 months) after transplantation and is the leading cause of death of transplanted patients. The pathogenesis of Chronic GVHD is still little known. Chronic GVHD is caused by donor T lymphocytes, but we have no precise knowledge on the participation of specific subsets of immune system cells to chronic GVHD. In general, chronic GVHD is associated with an increase in the number of T effector lymphocytes, both helper type 2 and cytotoxic.

Recently, also antigen presenting cells (APCs) have been implicated in pathogenesis of chronic GVHD in studies performed on animal models. T lymphocyte responses that characterize chronic GVHD require that recipient antigens are submitted by APCs which originate from the donor's HSC ( Hematopoietic Stem Cells) APCs are heterogeneous population that includes dendritic cells (DCs) ,monocytes, activated B lymphocytes and CD34+ cell subpopulations. These cells can be identified by cytometry.

The data about APCs role in chronic GVHD are preliminary and often discordant. Seemingly, there isn't correlation between circulating APCs number and risk of cGVHD. However, recent data of our group show that patients with cGVHD could have higher number of monocytes in bone marrow than transplanted patients without cGVHD.

The aim of study is to measure the number of circulating immune cells in the PB (peripherical blood) before and after Allogeneic Hematopoietic Stem Cell Transplantation by flow cytometry.

DETAILED DESCRIPTION:
Study Endpoints

The primary endpoint of study is detection of circulating cells by flow cytometry before and after Allogeneic Stem Cell Transplantation. We analyze the following cells: Myeloid Dendritic Cells, Plasmacytoid Dendritic cells, CD16+ Dendritic cells, CD14+ monocytes, CD14+/CD16+ monocytes, total T lymphocytes, total T helper lymphocytes, central memory, naive, effector memory and effector T helper lymphocytes, total cytotoxic lymphocytes, central memory, naive, effector memory and effector T cytotoxic lymphocytes, CD16+/CD56+ NK cells, B lymphocytes, T regulatory lymphocytes.

The secondary endpoints are:

* Determination of the serum concentration of Cytokines (TNFα, IFNγ, IL-4) and Chemokines ( MIP and MCP group).
* Determination of autoantibodies in the serum. In the first phase, screening analysis is performed by searching anti nuclear antibodies (ANA) and antibodies anti-ENA (Extractable Nuclear Antigens). Positive results are subjected to second level analysis. Next, we are proceed to the analysis of different Organ-Specific Autoantibodies, previously associated with chronic GVHD, like liver antibodies (SMA, AMA, SLA), anti-cardiolipin and beta2 microglobulin antibodies, Antibodies against thyroid and gastric parietal cells.
* Study of CD86, CXCR4, CCR2, CCR5, CD11a and CD49d molecules expression in Monocytes and Dendritic Cells.
* Study of TNF and IL-12 production by purified monocytes
* Study of Allostimulatory activity of purified monocytes against Allogeneic CD4+ T cells.
* Study of antigen capture and processing by phagocytosis, macropinocytosis and endocytosis mediated by purified monocytes receptors.
* Study of CD134 (0X40L), CD154 (CD40L) molecules expression, study of differentiation molecules type1 and type 2 T helper cells and T regulatory Cells associated, study of molecules Cellular Death associated.
* Study of Cytokines proliferation and production (including IL-2, IL-5, IFNγ and IL-10) and release of perforin and granzyme after stimulation with mitogens.
* Study of antigen-specific T lymphocytes response by pentamers for detection of HY antigen by ELISPOT assay. Recipient's cells are collected and stored before the transplantation
* PCR study of micro (mi) RNA in patient's serum and cells.
* PCR and Microarray study of gene expression profile of transplanted monocytes

Study design

Observational single center prospective study employing human tissues for in vitro study after Allogeneic Stem Cell Transplantation. The study includes a retrospective phase. The study requires that patient's Peripheral blood samples are harvested :

* on entering the department
* after 1 month of transplantation
* after 3, 6, 9,12 months of transplantation

Study Population

All patients undergoing Allogeneic Transplantation in our Institute are included.

Collection and processing of blood samples

Each peripheral blood sample must be collected in three heparin tubes ( up to 18 ml of SP) and a non-anticoagulant tube (6 ml for a total of at least 3 ml of serum)

Each sample is processed as follows:

Blood sample taken without anticoagulant will be centrifuged to obtain serum, the aliquots of serum are frozen and stored at -20°C The immunophenotypic analysis for number and function of the mentioned cells are performed on fresh PB samples within 72 hours of collection.

Mononuclear cells and monocytes are purified by standard procedures (MNCs by density gradient centrifugation, monocytes by immunomagnetic selection) and then stored in liquid nitrogen until they are used for expected functional assays. The negative CD14 fraction are frozen and used as the source of T lymphocytes.

Flow cytometry analysis

The number and phenotype of the immune system circulating cells are determinated by flow cytometry using the specific monoclonal antibodies.We are considered the following immune cells :

* CD4+ and CD8+ T lymphocytes including T naïve lymphocytes (CD45RA + CCR7 +) "effector" memory lymphocytes (CD45RA-CCR7-), "central" memory lymphocytes (CD45RA-CCR7 +) and effector lymphocytes (CD45RA-CCR7 +).
* T regulatory lymphocytes (CD4 + CD25 + CD127-FoxP3 +).
* B Lymphocytes (CD19 +)
* NK cells (CD56 + CD16-) and cytotoxic (CD56 + CD16 +) cells.
* Myeloid Dendritic Cells CD11c + (lineage-, DR +, CD33 +), Plasmacytoid Dendritic Cells (lineage-, DR +, CD33- and CD123 +) and Monocytoid (CD33 +, CD14-, CD16 +) DCs.
* Inflammatory (CD14 + CD16 +) and Constituents (CD14 + CD16-) Monocytes

Functional studies on purified monocytes

* TNF alpha and IL12 production are measured in flow cytometry.
* The allostimulatory function is determined in mixed leukocyte cultures using HLA different CD4 + T lymphocytes as "responders".
* The ability to capture antigens is measured in flow cytometry on individual cells by fluorescence antigens, such as FITC conjugated albumin or fluorescent beads.
* The gene expression profile is performed using a MICROARRAY study

Functional studies on purified T lymphocytes

* The expression of activation, differentiation and apoptosis molecules is determinated by cytometry
* Cytokine production is determined in single-color flow cytometry after stimulation with anti-CD3 and anti-CD28.
* In positive male HLA-A2 patients receiving female donor transplantation, the frequency of T anti-HY lymphocytes is measured by fluorochrome-conjugated pentamers.
* In all other patients, T-cell donor response to receptor antigens is measured in ELISPOT.

Serum cytokines Study

The concentration of serum cytokines is determined in cytometry using CBA (Cytokine Bead Assay, CBA, Becton Dickinson, Mountian View, CA, USA). We analyze the following cytokines:

* T-helper 1 cytokines: TNF-alpha, IFN-gamma and IL-12;
* T-helper 2 and regulators cytokines (IL-10, IL-5), and TGF-beta
* Chemokines: MCP1, MCP2, RANTES, MIP1-alpha and MIP1-beta; IL-8, IP-10.

Serum autoantibodies Study

The concentration of the antinuclear antibodies is measured by indirect immunofluorescence on HEp2 cells (a cell line of hepatocarcinoma). The antibodies against extractable nuclear antigens (ENA) are measured by ELISA (ENA SCREENING). In case of positivity, the presence of antibodies against specific antigens is determined by DOT BLOT.

micro(mi) RNA PCR study in patient's serum and cells

The total RNA is extracted from human serum samples and stored at -80 ° C. A part of RNA ( 3µl) is processed for reverse transcription and pre-amplification with a pool of primers according to the supplier's description. 664 human miRNA, 6 small human RNA and 1 control miRNA are processed in parallel.

Gene expression profile Study of transplanted patient's monocytes by PCR and MICROARRAY

The monocyte RNA messenger is extracted from the cells, converted into cDNA by reverse transcriptase and at the same time labeled with a fluorescent probe. The hybridization between the nucleic acids (probes) present on the matrix and the cDNA target will remain hybridized and can then be identified by detecting the location where it is bound. At the end of study, all samples will be destroyed.

Concomitant treatments

Patients will receive or have received chemotherapy for transplant preparation according to current clinical practice. After transplantation, patients will receive medication for prophylaxis of GVHD and infections according to clinical practice. Concomitant therapies possibly administered according to clinical practice are documented in CRF.

Schedule of visits and evaluations

Patient visit is expected and CRF is completed at the enrollment. There are 6 blood samples per patient. Any blood sample after the enrollment can be delayed or anticipated by 14 days

Laboratory Tests

Tests are performed under the normal care pathway and are not study-specific. Blood exam informations are reported on CRFs.

Statistical analysis

The primary endpoint of the study is the measure of circulating immune cell number in PB before and after Allogeneic Hematopoietic Stem Cell Transplantation. Statistical analysis consists of comparison analysis between averages using GRAPH PAD PRISM version 4.02 program. The level of significance is defined as <.05 Analysis of secondary endpoints is performed using the same methods.

Sample Size

The study is proposed to all patients undergoing allogeneic transplantation. The number of transplants performed at the Seràgnoli Institute is on average between 50 and 60 per year. It is therefore estimated that 300 patients will be enrolled in the study.

Administrative procedures

Any modification to the protocol will be made in the form of the amendment. No other types of modification to the protocol are allowed during the study period. Any unexpected changes in the study will be recorded in the Clinical Study Report.

Management of informed consent

All patients date and write the Informed Consent within one of the visits provided by the normal care path. For dead patients, it is considered that the data processing is authorized with the approval of the study by the Ethics Committee, according to general authorization (Official Journal 72 of 26/03/2012)

Documentation archive

The principal Investigator is responsible for storing of the essential documents of the study before, during, and after the completion or termination of the study, in accordance with the time required by the applicable laws and GCPs.

The data collected in the CRF are strictly anonymous and the subject is only identified with a number and initials.

The Investigator will have to keep the patient's original data and informed written consent.

Inspections / Audits

If a Regulatory Authority requires an inspection, the Investigator must immediately inform the Ethics Committee.

Publication of results

The results of the experiment will be published within twelve months of the conclusion.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing Allogeneic hemapoietic Stem Cell Transplantation

Exclusion Criteria:

Patient not undergoing allogeneic hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing Allogeneic Stem Cell Transplantation are enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of study is detection of circulating cells by flow cytometry before and after Allogeneic Stem Cell Transplantation | Patient's PB samples are harvested : on entering the department;1 month after transplantation ; 3, 6, 9,12 months after transplantation
  We analyze the following cells:Myeloid Dendritic Cells, Plasmacytoid Dendritic cells, CD16+ Dendritic cells, CD14+ monocytes, CD14+/CD16+ monocytes, total T lymphocytes, total T helper lymphocytes, central memory, naive, effector memory and effector T helper lymphocytes, total cytotoxic lymphocytes, central memory, naive, effector memory and effector cytotoxic lymphocytes, CD16+/CD56+ NK cells, B lymphocytes, T regulatory lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Arpinati, MD, Principal Investigator — St. Orsola-Malpighi University Hospital Bologna, Italy
Locations (1):
- Mario Arpinati, Bologna, Italy

REFERENCES:
- [Background] Nakamura K, Amakawa R, Takebayashi M, Son Y, Miyaji M, Tajima K, Nakai K, Ito T, Matsumoto N, Zen K, Kishimoto Y, Fukuhara S. IL-4-producing CD8(+) T cells may be an immunological hallmark of chronic GVHD. Bone Marrow Transplant. 2005 Oct;36(7):639-47. doi: 10.1038/sj.bmt.1705107. PMID 16044136
- [Background] D' Asaro M, Salerno A, Dieli F, Caccamo N. Analysis of memory and effector CD8+ T cell subsets in chronic graft-versus-host disease. Int J Immunopathol Pharmacol. 2009 Jan-Mar;22(1):195-205. doi: 10.1177/039463200902200122. PMID 19309567
- [Background] Arpinati M, Chirumbolo G, Saunthararajah Y, Stanzani M, Bonifazi F, Bandini G, Baccarani M, Rondelli D. Higher numbers of blood CD14+ cells before starting conditioning regimen correlate with greater risk of acute graft-versus-host disease in allogeneic stem cell transplantation from related donors. Biol Blood Marrow Transplant. 2007 Feb;13(2):228-34. doi: 10.1016/j.bbmt.2006.10.004. PMID 17241928
- [Background] Anderson BE, McNiff JM, Jain D, Blazar BR, Shlomchik WD, Shlomchik MJ. Distinct roles for donor- and host-derived antigen-presenting cells and costimulatory molecules in murine chronic graft-versus-host disease: requirements depend on target organ. Blood. 2005 Mar 1;105(5):2227-34. doi: 10.1182/blood-2004-08-3032. Epub 2004 Nov 2. PMID 15522961
- [Background] Arpinati M, Chirumbolo G, Marzocchi G, Baccarani M, Rondelli D. Increased donor CD86+CD14+ cells in the bone marrow and peripheral blood of patients with chronic graft-versus-host disease. Transplantation. 2008 Jun 27;85(12):1826-32. doi: 10.1097/TP.0b013e3181788a84. PMID 18580477